CLINICAL TRIAL: NCT02200536
Title: Effectiveness of an Oral Health Promotion Program in Infant's Tooth Brushing and Bottle-feeding Termination Practices: a Randomized Controlled Trial
Brief Title: Impact of Providing Free Preventive Dental Health Products on Infant's Tooth Brushing and Bottle-feeding Termination Practices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DM20AM18
Record Dates: First submitted 2014-07-22; First posted 2014-07-25 (Estimated); Results first posted 2015-03-27 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Infant's Tooth Brushing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Test (Experimental): Infant oral health promotion package
  Interventions: Other: Infant oral health promotion package
- Control 1 (Active Comparator): Infant oral health pamphlet
  Interventions: Other: Infant oral health pamphlet
- Control 2 (No Intervention)

INTERVENTIONS:
Other: Infant oral health promotion package — Infant oral health promotion package includes an infant oral health pamphlet, a baby toothbrush, fluoride toothpaste (1000 ppm) and a trainer cup.
  Arms: Test
Other: Infant oral health pamphlet — Infant oral health pamphlet
  Arms: Control 1

SUMMARY:
Governmental initiatives (such as Sure Start in the UK) have integrated an oral health promotion intervention within their maternal and child health program and delivered dental education and enabling resources (a gift bag including a baby toothbrush, fluoride toothpaste and a trainer cup) to infant's mothers. Whilst this approach has minimal financial implications of human resources, no evidence exists regarding its effectiveness in establishing desirable infant's oral health behaviours. In Syria, there is a great need for developing an infant's oral health promotion program to promote oral hygiene practice, provide access to fluoride and terminate bottle-feeding practice. Thus, the current study aimed to test the effectiveness of an integrated infant's oral health promotion intervention within the Syrian national immunization program, which delivered printed dental education materials, a baby tooth brush, fluoride toothpaste (1000 ppm) and a trainer cup, in establishing one-year old infant's oral hygiene and bottle-feeing termination practices.

DETAILED DESCRIPTION:
The current randomized controlled trail allocated 92 one-year old infants, attending a maternal and child health center in Sweida city-Syria, to receive their vaccination, into three groups: test, control 1 and control 2. The test group received an infant oral health promotion package including a child oral health pamphlet, a baby toothbrush, fluoride toothpaste (1000 ppm) and a trainer cup. Control 1 received only an infant pamphlet, whilst Control 2 received no intervention. A mother's self-completed structured questionnaire and an infant's clinical examination were completed and performed, at baseline and after one month, to assess tooth brushing and bottle-feeding practices as well as the presence of old plaque on infant's primary teeth, respectively.

ELIGIBILITY:
Inclusion Criteria for infants:

* Healthy
* Single (not twins).
* Full-term (≥37 weeks).
* Birth weight ≥ 2500 g.
* Family size ≤3 children (including the infant).
* Their first tooth erupted.
* No reported tooth brushing practice.

Ages: 12 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2013-03; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Easter Joury, BDS, DOrth, MSc, PhD, Study Director — Damascus Univeristy; Muna Alghadban, BDS, MSc, Principal Investigator — Damascus University
Locations (1):
- Faculty of Dentistry, Damascus, Syria

RESULTS

PARTICIPANT FLOW:
Groups:
- Control 2: No intervention.
Period: Overall Study
Arm/Group | Test | Control 1 | Control 2
Started | 32 | 30 | 30
Completed | 32 | 30 | 30
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test | Control 1 | Control 2 | Total
Number analyzed (Participants) | 32 | 30 | 30 | 92
Age, Customized [Number; unit: participants] — Mother's age
  participants
    ≥ 30 years old | 11 | 16 | 17 | 44
    < 30 years old | 21 | 14 | 13 | 48
Sex: Female, Male [Count of Participants; unit: Participants] — Infant's gender, Male/Female
  Participants
    Female | 19 | 21 | 19 | 59
    Male | 13 | 9 | 11 | 33

OUTCOME MEASURES:

1. Primary Outcome: Change in Mother's Reported Infant's Twice-a-day Tooth Brushing Practice.
Description: Change in mother's reported infant's twice-a-day tooth brushing practice was measured by comparing mother's reported infant's twice-a-day tooth brushing practice at follow up and baseline. Change was present when mother's reported infant's twice-a-day tooth brushing practice after one month compared to mother's reported no infant's twice-a-day tooth brushing practice at baseline. Change was not present when mother's did not report infant's twice-a-day tooth brushing practice after one month compared to mother's reported no infant's twice-a-day tooth brushing practice at baseline.
Time Frame: Baseline (T0) and after one month (T1)
Measure: Number; unit: percentage of mothers
Arm/Group | Test | Control 1 | Control 2
Number analyzed (Participants) | 32 | 30 | 30
percentage of mothers | 90.6 | 10 | 6.7

2. Secondary Outcome: Change in Mother's Reported Bottle-feeding Practice.
Description: Change in mother's reported bottle-feeding practice was measured by comparing mother's reported bottle-feeding practice at follow up and baseline. Change was present when mother's reported no bottle-feeding practice after one month compared to mother's reported bottle-feeding practice at baseline. Change was not present when mother's reported bottle-feeding practice after one month compared to mother's reported bottle-feeding practice at baseline.
Time Frame: Baseline (T0) and after one month (T1)
Measure: Number; unit: percentage of mothers
Arm/Group | Test | Control 1 | Control 2
Number analyzed (Participants) | 16 | 13 | 16
percentage of mothers | 18.8 | 69.2 | 93.8

ADVERSE EVENTS:
Description: Serious or other [non-serious] adverse events were not collected in the current trial, as there were no previously identified adverse events in studies with the same type of interventions.
Arm/Group | Test | Control 1 | Control 2
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No